CLINICAL TRIAL: NCT07157904
Title: Evaluating the PATHFAST TB LAM Ag Assay as a Treatment Monitoring Tool for Pulmonary Tuberculosis: A Prospective Longitudinal Study in Nairobi, Kenya
Brief Title: Evaluation of PATHFAST-LAM as a Tuberculosis Treatment Monitoring Tool in Kenya
Status: Not yet recruiting | Type: Observational
Sponsor: Nagasaki University (Other)
Responsible Party: Principal Investigator, Nobuo Saito, Associate Professor, Nagasaki University
Other Study IDs: KEMRI/SERU/CRDR/124/5241
Record Dates: First submitted 2025-08-28; First posted 2025-09-05 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Tuberculosis; Pulmonary Tuberculoses; Mycobacterium Tuberculosis
Keywords: Tuberculosis; Treatment Monitoring Tool; Lipoarabinomannan
MeSH Terms: conditions — Tuberculosis; Tuberculosis, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pulmonary Tuberculosis Patients

SUMMARY:
Tuberculosis (TB) can be treated; however, the standard 6-month treatment is long and challenging for many patients, and 10-20% still don't recover well by the end of treatment. Thus, it's important to regularly check if the treatment is working to help patients get better and prevent drug-resistant TB from developing. It can, however, be especially hard to check if TB treatment is working in places with limited resources. Traditional methods, such as testing sputum samples for microscopy and culture, have limitations. Lipoarabinomannan (LAM) is a substance that is found in the cell wall of the bacteria that cause TB, which can be used as an indicator for TB diagnosis and treatment monitoring. The PATHFAST TB LAM Ag test is a fully automatic machine that checks for LAM in sputum. It could offer a faster and more accurate way to see if TB treatment is working. This study aims to find out how helpful the PATHFAST-LAM test is in monitoring TB treatment progress among Kenyan TB patients.

The primary objective of this study is to assess whether changes in sputum LAM levels can help predict unfavorable results.

In this study, investigators will recruit adult patients diagnosed with pulmonary TB from multiple healthcare facilities in Nairobi, Kenya. Investigators will follow them during their TB treatment and collect sputum and urine samples at the beginning of treatment, then, every week for the first month, every two weeks for the next two months, and monthly for months 3-6. Investigators will use the PATHFAST-LAM test to measure LAM levels in sputum and urine. Since there are no previous studies that have evaluated the relationship between sputum LAM and treatment outcome, investigators will do an initial analysis with 30 participants, and based on that, investigators will determine the final number of participants needed for our study.

It is expected that sputum LAM decreases when the treatment is successful and remains positive (does not decrease) when treatment is unsuccessful, with patients experiencing unfavorable results. How LAM decreases during the earlier course of TB treatment may be useful in predicting patients' outcomes. The results of this study could provide a faster and effective way for monitoring TB treatment. This could contribute to improved patient outcomes and help reduce the global burden of TB.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Patients with a recent diagnosis of bacteriologically confirmed PTB who have not yet initiated TB treatment.
* Patients who are willing and able to visit to the facility for follow-up sample collection and interviews.
* Patients who are willing and able to provide written informed consent to participate in the study.

Exclusion Criteria:

- Patients with a history of TB treatment within the past 6 months, including retreatment.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: To ensure a representative sample reflecting a broad spectrum of TB disease severity and healthcare access, investigators will recruit participants from multiple healthcare facilities at different levels of the Kenyan health system. The primary study sites include Rhodes Chest Clinic (RCC) and Mbagathi County Referral Hospital (MCH). RCC is a Level 2 healthcare facility which serves as a specialized primary care center for TB patients, recording approximately 700-800 new PTB cases every year. MCH is a Level 5 referral hospital offering both outpatient and inpatient care with a bed capacity of around 150. MCH manages 1,000 new TB cases annually.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Composite Poor Outcome | From enrollment to 3 months after treatment completion
  Patients who meet any of the following criteria: (1) Death due to any cause, (2) Discontinuation of TB treatment for more than 2 months consecutively, (3) Early relapse (within 3 months after completing TB treatment), (4) Change in TB treatment regimen for any reason, or (5) No culture conversion at the end of TB treatment.

CONTACTS AND LOCATIONS:
Locations (2):
- Kenya (2):
  - Mbagathi County Referral Hospital, Nairobi
  - Rhodes Chest Clinic, Nairobi

REFERENCES:
- [Derived] Takaizumi Y, Kinoti J, Hikone M, Orina F, Meme H, Ong'ang'o JR, Muriithi B, Mueni E, Kaneko S, MacLean EL, Sato S, Saito N. Evaluating the PATHFAST TB LAM Ag assay as a treatment monitoring tool for pulmonary tuberculosis: protocol for a prospective longitudinal study in Nairobi, Kenya. BMJ Open. 2026 Jan 13;16(1):e113578. doi: 10.1136/bmjopen-2025-113578. PMID 41529882